CLINICAL TRIAL: NCT00210483
Title: A Randomized, Double-blind, Placebo-controlled Study of Oral Almotriptan Malate (AXERT®) 6.25 mg, 12.5 mg, and 25 mg in the Acute Treatment of Migraine in Adolescents
Brief Title: A Study of 3 Dosage Strengths of Almotriptan Malate (AXERT®) in the Treatment of Acute Migraine in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho LLC (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004567
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Migraine
Keywords: pain; Migraine; aura; headache
MeSH Terms: conditions — Migraine Disorders; Pain; Epilepsy; Headache | interventions — almotriptan

INTERVENTIONS:
Drug: almotriptan malate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of almotriptan malate (AXERT®) in treating acute migraine headaches in adolescents. Amotriptan malate (AXERT®) is approved for use in the treatment of acute migraine headache with or without aura in adults. In this study, adolescents will be given a single dose of study medication to treat one migraine headache.

DETAILED DESCRIPTION:
Amotriptan malate (AXERT®) is approved for use in the treatment of acute migraine headache with or without aura in adults. Other studies have shown that almotriptan is effective and well tolerated in adults. Migraines in teenagers/adolescents are very similar to migraines in adults, except that the duration is usually less in adolescents (they last 1 to 24 hours in adolescents). This study will evaluate the usefulness of almotriptan malate (AXERT®) in treating acute migraine headaches in adolescents. This is a randomized, double-blind, parallel-group, and placebo-controlled study. During a 30-day run-in period, patients will treat their migraines as they normally would. During this time, the frequency and severity of headaches will be recorded. At the second visit, patients will be randomized (like with the toss of a coin) to a treatment group to receive one oral dose of almotriptan malate (AXERT®) 6.25, 12.5, or 25 milligrams or placebo. Approximately the same number of patients will be assigned to each of the four treatment groups. Patients will take this one-time dose when the next migraine of at least moderate severity occurs. Patients will record assessments in a diary for up to 24 hours after the study drug is given to help determine the drug's effect on headache pain intensity. Patients will return for a third visit within 2 to 14 days from taking the study medication. A physical examination, electrocardiogram (a painless test of the heart), and laboratory tests will be performed at the first and third visits. The objective of this study is to determine the effectiveness and tolerability of 3 dosage strengths of almotriptan malate (AXERT®) in adolescents with migraine headaches.

Almotriptan oral tablets, 6.25, 12.5, or 25 milligrams, or placebo

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with or without aura for > 1 year
* Average of 1 to 6 moderate or severe migraines per month for 2 months before entering the study
* Untreated migraines lasting at least 4 hours
* At least 24 hours between migraines
* Able to tell the difference between migraines and other types of headache
* If female, using birth control

Exclusion Criteria:

* Chronic tension or cluster headache
* Prolonged aura
* Specific types of migraine
* > 6 nonmigraine headaches per month
* High blood pressure for the age
* Medical history with specific significant conditions affecting the liver, kidney, heart or other body systems
* Conditions that might affect the way the body absorbs or processes a drug
* Positive blood tests for Hepatitis B or C
* Recent head or neck injury
* Body weight outside given parameters
* Unable to take sumatriptan
* Abusing drugs or alcohol
* Pregnant or breast-feeding
* Use of antimigraine medication that might interfere with the study, of antimigraine medication for < 2 weeks, of lithium or monoamine oxidase inhibitors in past 2 weeks, of an investigational drug within 2 months
* Refuse to abstain from taking medicine with ergotamine or any other drug like almotriptan within 48 hours before and 24 hours after taking study medication, or drugs containing opiates or antivomiting medicine within 48 hours before and 2 hours after taking study medication
* Use of simple pain medicines within 24 hours (like aspirin)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 866 (Actual)
Dates: Start 2003-07; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Efficacy determined by patient 2 hours after dosing by rating of headache intensity as a decrease from moderate or severe to mild or no pain

SECONDARY OUTCOMES:
Efficacy, symptoms, headache pain free at time points 0.25, 0.5, 1, 1.5 hours postdose; incidence of headache recurrence in 2 to 24 hours and use of rescue medication 2 to 24 hours postdose; pain relief or pain free at 24 hours; all by patient assessment

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Ortho LLC Clinical Trial, Study Director — Janssen-Ortho LLC

REFERENCES:
- [Derived] Linder SL, Mathew NT, Cady RK, Finlayson G, Ishkanian G, Lewis DW. Efficacy and tolerability of almotriptan in adolescents: a randomized, double-blind, placebo-controlled trial. Headache. 2008 Oct;48(9):1326-36. doi: 10.1111/j.1526-4610.2008.01138.x. Epub 2008 May 14. PMID 18484981
- See also: Axert in Pediatric Migraine — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=292&filename=CR004567_CSR.pdf